CLINICAL TRIAL: NCT05678582
Title: The Impact of Hepatic Steatosis on Chronic Hepatitis B Virus Infection
Brief Title: Hepatic Steatosis and Chronic Hepatitis B Virus
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mona Mohammed Abdelrhman, Principal investigator, Sohag University
Other Study IDs: Soh-Med-22-12-26
Record Dates: First submitted 2022-12-19; First posted 2023-01-10 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Chronic Hepatitis
Keywords: HBV; Steatosis
MeSH Terms: conditions — Hepatitis, Chronic; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Ultrasound-guided percutaneous liver biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HBV with hepatic steatosis: HBV with hepatic steatosis on liver biopsy
  Interventions: Diagnostic Test: Liver biopsy
- HBV without hepatic steatosis: HBV without hepatic steatosis on liver biopsy
  Interventions: Diagnostic Test: Liver biopsy

INTERVENTIONS:
Diagnostic Test: Liver biopsy — liver biopsy were taken then evaluated by histopathological examination

SUMMARY:
This study aims to evaluate the prevalence and severity of hepatic steatosis in CHB and investigate the relationship between hepatic steatosis and viral load, liver biochemistry, liver fibrosis, and inflammation in CHB

DETAILED DESCRIPTION:
This hospital-based cohort study will be conducted on 80 adult hepatitis B surface antigen (HBsAg) carriers presented to the Tropical Medicine and Gastroenterology outpatient clinic, at Sohag University Hospital Exclusion criteria Patients with serological evidence of HCV. HBV patients who had received or are currently under anti-viral therapy. Alcohol consumption. Decompensated liver disease. Patients with HCC. Patients are known to have another chronic liver disease (e.g. autoimmune hepatitis, primary biliary cirrhosis, Wilson's disease, Haemochromatosis, or drug-induced chronic hepatitis).

Patients with contraindications to liver biopsy such as uncooperative patients, prothrombin time (PT) >4 seconds more than control, INR greater than 1.6, platelets count <100.000/mm3After taking informed written consent, the participants will be subjected to:

Clinical evaluation: medical history and physical examination.

Laboratory investigations:

Complete blood count. Prothrombin time and concentration. Liver function tests Anti-HCV. HBeAg. HBV DNA. Abdominal ultrasonography Ultrasound-guided percutaneous liver biopsy

ELIGIBILITY:
Inclusion Criteria:

Hepatitis B surface antigen (HBsAg) carriers presented to the Tropical Medicine and Gastroenterology outpatient clinic, at Sohag University Hospital

Exclusion Criteria:

Patients with serological evidence of HCV. HBV patients who had received or are currently under anti-viral therapy. Alcohol consumption. Decompensated liver disease. Patients with HCC. Patients are known to have another chronic liver disease (e.g. autoimmune hepatitis, primary biliary cirrhosis, Wilson's disease, Haemochromatosis, or drug-induced chronic hepatitis).

Patients with contraindications to liver biopsy such as uncooperative patients, prothrombin time (PT) >4 seconds more than control, INR greater than 1.6, platelets count <100.000/mm3.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 91 adult Hepatitis B surface antigen (HBsAg) carriers presented to the Tropical Medicine and Gastroenterology outpatient clinic, at Sohag University Hospital.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
prevalence of hepatic steatosis in CHB | January 2023 to july 2023 will be included in the study
  Number of cases with hepatic steotosis in CHB
degree of hepatic steatosis in CHB | January 2023 to july 2023 will be included in the study
  Mild, or Moderate or severe degree

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa Sadek, MD, Study Chair — Sohag University
Locations (1):
- Faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365
- [Background] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875